CLINICAL TRIAL: NCT01153516
Title: Unraveling the Mechanisms of Rapid Improvement in Diabetes Following Gastric By-Pass Surgery
Brief Title: Diabetes and Gastric By- Pass
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ildiko Lingvay, MD, MPH, MSCS, University of Texas Southwestern Medical Center
Other Study IDs: 122009-049
Record Dates: First submitted 2010-06-24; First posted 2010-06-30 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Bariatric surgery; Obesity; Weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood samples, plasma, serum, urine,
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the mechanisms leading to rapid postoperative improvement in diabetes following Gastric By-Pass surgery for obesity.We will evaluate and compare the changes in glucose level, beta-cell function, and insulin resistance induced by a week of very low calorie liquid diet and those induced by a week of matched very -low calorie liquid diet occuring in the context of routine postoperative care following RYGB.

DETAILED DESCRIPTION:
Volunteers planned to undergo RYGB will be studied during two-9 days periods of identical and controlled diet and activity, separated by a 4-10-week washout period.

Study Period #1:

This first study period is 9 days/nights long and requires you to be closely supervised at our Clinical and Translational Research Center (CTRC). During this time you will receive the same diet and are expected to have the same activity level you will be prescribed in the immediate post-operative period.

Wash-out period:

During this study period you are expected to return to your usual diet and exercise level.

Study Period #2:

This last study period is also 9 days/nights long, includes the EXACT same diet you have received during the first study period, and in addition you will undergo the planned gastric by-pass surgery.

Procedures during the research:

Mixed Meal Challenge test will be done four times during the entire study: days 1 and 9 for each study period. This test allows the investigators to evaluate how much insulin your body is producing and how well this insulin is processed.

Measurement of resting energy expenditure will be done four times during the entire study. This test tell us how much energy your body is burning up in a resting state.

ELIGIBILITY:
Inclusion Criteria:

* volunteers that are planned to undergo RYGB(Roux-en-Y By pass) and have type 2 diabetes diagnosed within the prior 10 years.

Exclusion Criteria:

* abnormal renal function
* significant anemia
* difficult venous access
* treatment with incretin mimetics or DPP IV inhibitors in the prior 3 months
* recent change in use of any pharmacologic agent with potential effect on either beta-cell function or insulin resistance.
* pregnancy
* non -English speakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bariatric surgery clinical roster or by the treating physician in the bariatric surgery clinic.
  This study does NOT pay for the By-pass surgery, eligible participants should have planned their surgery by their own physician, at their own expense.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Lingvay, MD, MPH, MSCS, Principal Investigator — UT Southwestern Medical Center, Dallas
Locations (1):
- Clinical and Translational Research Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Lingvay I, Guth E, Islam A, Livingston E. Rapid improvement in diabetes after gastric bypass surgery: is it the diet or surgery? Diabetes Care. 2013 Sep;36(9):2741-7. doi: 10.2337/dc12-2316. Epub 2013 Mar 25. PMID 23530013

RESULTS

PARTICIPANT FLOW:
Groups:
- Diet Only Group: Patients on diet and activity protocol typical for patients after bariatric surgery
- Surgery and Diet Group: Patients on diet and activity protocol typical for patients after bariatric surgery followed by Roux-en-Y gastric bypass surgery.
Period: Overall Study
Arm/Group | Diet Only Group | Surgery and Diet Group
Started | 12 | 10
Completed | 10 | 10
Not Completed | 2 | 0
Not completed — Both subjects refused surgery | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Only Group | Surgery and Diet Group | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (8.1) | 53.2 (8.4) | 53.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Response in Glucose AUC at Baseline vs. Following Gastric Bypass Surgery
Description: Changes in the glucose Area Under the Curve (AUC) calculated as the difference between the initial evaluation (test 1, assessed at day 1) and the next evaluation (test 2, assessed at day 9) of study period 1. Subjects then underwent gastric bypass surgery approximately 4-10 weeks later. In study period 2 following surgery, changes in the glucose AUC was again calculated as the difference between the initial evaluation (test 3, assessed at day 1 following surgery) and the next evaluation (test 4, assessed at day 9 following surgery). Change in AUC in study period 1 was compared to change in AUC in study period 2.
  Blood samples were collected at 5, 10, 15, 20, 25, 30, 40, 50, 60, 80, 100, 120, 150, 180, 210, 240, 300, and 360 minutes after the ingestion of 240 mL of chocolate Boost Plus Nestle.
  Total AUC was computed using the trapezoidal rule.
Time Frame: 4-12 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL*min
Arm/Group | Diet Only Group | Surgery and Diet Group
Number analyzed (Participants) | 10 | 10
mg/dL*min | 61647.0 [47023.3 to 76270.8] | 59476.1 [47943.8 to 71008.4]

2. Primary Outcome: Response in Insulin AUC at Baseline vs Following Gastric Bypass Surgery
Description: Changes in the Insulin Area Under the Curve (AUC) calculated as the difference between the initial evaluation (test 1, assessed at day 1) and the next evaluation (test 2, assessed at day 9) of study period 1. Subjects then underwent gastric bypass surgery approximately 4-10 weeks later. In study period 2 following surgery, changes in the insulin AUC was again calculated as the difference between the initial evaluation (test 3, assessed at day 1 following surgery) and the next evaluation (test 4, assessed at day 9 following surgery). Change in AUC in study period 1 was compared to change in AUC in study period 2.
  Blood samples were collected at 5, 10, 15, 20, 25, 30, 40, 50, 60, 80, 100, 120, 150, 180, 210, 240, 300, and 360 minutes after the ingestion of 240 mL of chocolate Boost Plus Nestle.
  Total AUC was computed using the trapezoidal rule.
Time Frame: 4-12 weeks
Measure: Mean (95% Confidence Interval); unit: uIU/mL*min
Arm/Group | Diet Only Group | Surgery and Diet Group
Number analyzed (Participants) | 10 | 10
uIU/mL*min | 7888.6 [5505.19 to 10272.08] | 4259.3 [3262.1 to 5256.4]

3. Primary Outcome: Response in Glucagon AUC at Baseline vs. Following Gastric Bypass
Description: Changes in the glucagon Area Under the Curve (AUC) calculated as the difference between the initial evaluation (test 1, assessed at day 1) and the next evaluation (test 2, assessed at day 9) of study period 1. Subjects then underwent gastric bypass surgery approximately 4-10 weeks later. In study period 2 following surgery, changes in the glucagon AUC was again calculated as the difference between the initial evaluation (test 3, assessed at day 1 following surgery) and the next evaluation (test 4, assessed at day 9 following surgery). Change in AUC in study period 1 was compared to change in AUC in study period 2.
  Blood samples were collected at 5, 10, 15, 20, 25, 30, 40, 50, 60, 80, 100, 120, 150, 180, 210, 240, 300, and 360 minutes after the ingestion of 240 mL of chocolate Boost Plus Nestle.
  Total AUC was computed using the trapezoidal rule.
Time Frame: 4-12 weeks
Measure: Mean (95% Confidence Interval); unit: pg/mL*min
Arm/Group | Diet Only Group | Surgery and Diet Group
Number analyzed (Participants) | 10 | 10
pg/mL*min | 24332.8 [20624.3 to 28041.3] | 32929.1 [25920.5 to 39937.8]

ADVERSE EVENTS:
Time Frame: 18 days
Arm/Group | Diet Only Group | Surgery and Diet Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 1/12 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diet Only Group (N=12) | Surgery and Diet Group (N=10)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No